CLINICAL TRIAL: NCT07041931
Title: Empowering Newcomer VOICES by Implementing and Evaluating a Trauma- Informed and Gender-responsive Group Intervention in School and School-based Health Center Sites
Brief Title: Empowering Newcomer Voices: A Trauma-Informed, Gender-Responsive Group Intervention in Schools (VOCES-NUEVAS)
Acronym: VOCES-NUEVAS
Status: Not yet recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Oakland Unified School District (Unknown)
Responsible Party: Sponsor
Other Study IDs: 24-42289; 7500252 (Other Grant/Funding Number: University of California, San Francisco)
Record Dates: First submitted 2025-06-11; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Mental Health
Keywords: school-based care; mental wellness; identity development; group interventions
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- school 1: The first of 4 eligible Oakland Unified School District and/or school-based health center school sites recruited for this project.
- school 2: The second of 4 eligible Oakland Unified School District and/or school-based health center school sites recruited for this project.
- school 3: The third of 4 eligible Oakland Unified School District and/or school-based health center school sites recruited for this project.
- school 4: The fourth of 4 eligible Oakland Unified School District and/or school-based health center school sites recruited for this project.

SUMMARY:
The goal of this study is to see if VOCES-NUEVAS, a school-based program for newcomer girls from Latin America, is helpful and easy to use. The main questions the investigators want to answer are:

* Is VOCES-NUEVAS a good fit for newcomer girls in schools?
* Does it help improve their mental health and well-being?

Students who are already part of the VOCES-NUEVAS program at four school-based health centers will take short surveys before and after the program and give feedback after each session. The adults leading the program will also share their thoughts in group discussions or interviews. The results will help improve the program and prepare for a larger study in the future.

DETAILED DESCRIPTION:
The number of newcomer youth from Latin America entering the U.S. has surged recently, with border crossings reaching a 20-year high. These youth face mental and stress-related health challenges compared to their non-migrant peers, including higher trauma symptoms, substance use, and psychosocial issues. Culturally attuned, evidence-based interventions in trusted settings like schools and school-based health centers (SBHCs) could address these needs. VOICES-LITE, a gender and trauma-responsive intervention for adolescent female-identifying students, aligns well with these needs. After piloting VOICES-LITE in Spanish with newcomer youth, local partners found it feasible and acceptable. However, feedback indicated that further cultural adaptations are needed to better fit the specific context and population.

The investigators propose a hybrid effectiveness-implementation study to evaluate the culturally adapted intervention, VOCES-NUEVAS. This study will involve an open trial at four selected OUSD school/SBHC sites to assess the feasibility, acceptability, and effectiveness of the intervention, providing insights for further refinement ahead of a future R01 trial. The four participating sites will be selected from OUSD/SBHC locations that serve newcomer students (see attached site list), based on the availability of providers who are facilitating the VOCES-NUEVAS group and have agreed to participate in the research. Providers who are already scheduled to implement the intervention with newcomer students at these sites will be recruited for the study.

The investigators will assess whether the culturally adapted VOCES-NUEVAS manual and implementation guide used in schools sufficiently address the needs of newcomer students and their supporting providers. Students participating in the intervention at these sites will be recruited to participate in the current study. They will be asked to complete pre- and post-intervention questionnaires and provide session-by-session feedback to further improve the intervention. Both participating providers and students will also be asked to participate in a focus group or exit interview to provide additional feedback.

Results from the study will be shared with community stakeholders and used in future research, including a future R01 randomized-controlled trial to assess VOCES-NUEVAS's impact on newcomer students' mental health, substance use, and long-term outcomes. This future trial will be a separate IRB application from the current study.

ELIGIBILITY:
Inclusion Criteria (Youth):

* current students of an Oakland Unified School District (OUSD) and/or School-based Health Center (SBHC) middle or high school site
* Eligible and registered to participate in a VOCES NUEVAS group during the 2024-2025 or 2025-2026 school year

Exclusion Criteria (Youth):

* Not proficient in Spanish
* Unable to provide informed consent or assent
* Does not meet eligibility criteria to participate in VOCES-NUEVAS intervention
* Not enrolled as a middle or high school at an OUSD school/SBHC site.

Inclusion Criteria (Provider):

* aged 18 years old or older
* current social worker or school provider working at one of the eligible Oakland Unified School District and/or School-based Health Center middle or high school sites
* Facilitating a VOCES NUEVAS group during the 2024-2025 or 2025-2026 school year
* Eligible to deliver school services at OUSD school/school-based health center sites
* Previously trained on Voices-LITE curriculum
* proficient in English and Spanish

Exclusion Criteria (Provider):

* Not proficient in Spanish and/or English language
* Not previously trained on the Voices-LITE intervention
* Not approved to deliver the VOCES-NUEVAS intervention to students at OUSD schools/SBHC sites
* Not leading a VOCES-NUEVAS group at an OUSD school/SBHC site during the 2024-2025 school year.

Min Age: 12 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Eligible participants include young people of any sex assigned at birth or gender expression who relate to or identify with the experiences of girls and women in society today.
Study Population: Youth population: OUSD middle or high school students ages 12-18 years old that are interested in participating in the VOCES-NUEVAS group at an eligible OUSD/SBHC school site in Oakland, California.
  Provider population: OUSD Voices-LITE trained providers ages 18 years old or older, planning on running a VOCES-NUEVAS group at an eligible OUSD/SBHC school site in Oakland, California.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2026-08 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Youth Session Feedback Forms | Weekly for 8 weeks during the 8-week group intervention period
  Participants will complete this 8-question form immediately following completion of group session. Questions are related to overall impressions of the group, how useful the group was, and how connected they felt with other participants and facilitators, whether they would recommend the group to others, and then rating each session activity on a 5-point scale.
Provider Session Feedback Forms | Weekly for 8 weeks during the 8-week group intervention period
  Group providers will complete this 15-question form immediately following completion of group session. Questions are related to number of attendees, what activities were completed, impressions of group participant engagement and comprehension for each activity, and provider feedback on their most favorite part of group, least favorite, and parts of group that need modification.

SECONDARY OUTCOMES:
Demographics | Twice, once at baseline and once after the 8-week intervention period
  Participants will complete this 13-question form once at baseline and again following the 8-week intervention period. The Demographic measure will ask the participants questions related to their background (e.g. age, country of origin, languages spoken), history of migration and settlement, educational background, gender identity, and sexual orientation.
Coping with Acculturative Stress in American Schools (CASAS-A) | Twice, once at baseline and once after the 8-week intervention period
  Participants will complete this 18-question form once at baseline and again following the 8-week intervention period. The CASAS-A measure will ask the participants questions related to their experiences and emotions surrounding their acculturation experience in the United States.
Fears of Deportation | Twice, once at baseline and once after the 8-week intervention period
  Participants will complete this 6-question form once at baseline and again following the 8-week intervention period.The Fears of Deportation measure includes questions related to fear and engagement with law enforcement such as if their family members have avoided reporting crimes and how deportation concerns impact their behaviors.
CAGE Adapted to Include Drugs (CAGE-IAD) | Twice, once at baseline and once after the 8-week intervention period
  Participants will complete this 8-question form once at baseline and again following the 8-week intervention period. The CAGE-IAD measure will ask the participants questions related to concerning alcohol and drug usage.
Generalized Anxiety Disorder-7 (GAD-7) | Twice, once at baseline and once after the 8-week intervention period
  Participants will complete this 7-question form once at baseline and again following the 8-week intervention period.The GAD-7 measure will assess the severity of participants' anxiety.
Patient Health Questionnaire-9 (PHQ-9) | Twice, once at baseline and once after the 8-week intervention period
  Participants will complete this 9-question form once at baseline and again following the 8-week intervention period.The PHQ-9 measure will assess the severity of participants' depression.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren M Haack, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
Our study involves a vulnerable population and sensitive topics, making privacy and confidentiality our top priority. To prevent potential re-identification and uphold participant trust, we are not sharing individual participant data (IPD). Our consent process assured strict confidentiality, and sharing even de-identified data could pose risks. However, we welcome inquiries about aggregated results and methodology.

REFERENCES:
- [Background] Sidamon-Eristoff AE, Cohodes EM, Gee DG, Pena CJ. Trauma exposure and mental health outcomes among Central American and Mexican children held in immigration detention at the United States-Mexico border. Dev Psychobiol. 2022 Jan;64(1):e22227. doi: 10.1002/dev.22227. PMID 35050507
- [Background] Martinez-Donate AP, Verdecias N, Zhang X, Jesus Eduardo GF, Asadi-Gonzalez AA, Guendelman S, Amuedo-Dorantes C, Rangel G. Health Profile and Health Care Access of Mexican Migration Flows Traversing the Northern Border of Mexico. Med Care. 2020 May;58(5):474-482. doi: 10.1097/MLR.0000000000001300. PMID 32028523
- [Background] Almeida J, Johnson RM, Matsumoto A, Godette DC. Substance use, generation and time in the United States: the modifying role of gender for immigrant urban adolescents. Soc Sci Med. 2012 Dec;75(12):2069-75. doi: 10.1016/j.socscimed.2012.05.016. Epub 2012 Jun 7. PMID 22727651
- [Background] Cleary SD, Snead R, Dietz-Chavez D, Rivera I, Edberg MC. Immigrant Trauma and Mental Health Outcomes Among Latino Youth. J Immigr Minor Health. 2018 Oct;20(5):1053-1059. doi: 10.1007/s10903-017-0673-6. PMID 29139024
- [Background] Betancourt TS, Newnham EA, Birman D, Lee R, Ellis BH, Layne CM. Comparing Trauma Exposure, Mental Health Needs, and Service Utilization Across Clinical Samples of Refugee, Immigrant, and U.S.-Origin Children. J Trauma Stress. 2017 Jun;30(3):209-218. doi: 10.1002/jts.22186. Epub 2017 Jun 6. PMID 28585740
- [Background] Bailey CA, Widener K. The nexus between immigration status, policy, and proceedings, and mental health. Curr Opin Psychol. 2022 Oct;47:101411. doi: 10.1016/j.copsyc.2022.101411. Epub 2022 Jul 3. PMID 35914487